CLINICAL TRIAL: NCT03181256
Title: Early Detection of Lung Cancer in the Medically Underserved Population
Brief Title: Early Detection of Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Eric Grogan, Associate Professor of Thoracic Surgery, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 1730; NCI-2017-00889 (Registry Identifier: NCI, Clinical Trials Reporting Program); CA152662 (Other Grant/Funding Number: National Cancer Institute (EDRN))
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, nasal epithelium, buccal epithelium, blood, urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening: Patients are followed up at 1, 2, 3, 4, and 5 years and undergo collection of sputum, nasal epithelium, buccal epithelium, blood, and urine samples. Patients also undergo pulmonary function tests, chest CT, and review of medical records
  Interventions: Procedure: Biospecimen Collection; Procedure: Pulmonary Function Test; Procedure: Computed Tomography (CT); Other: Laboratory Biomarker

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of sputum
Procedure: Biospecimen collection — Undergo collection of nasal epithelium
Procedure: Biospecimen collection — Undergo collection of buccal epithelium
Procedure: Biospecimen collection — Undergo collection of blood
Procedure: Biospecimen collection — Undergo collection of urine
Procedure: Pulmonary Function Test — Undergo pulmonary function test
Procedure: Computed Tomography (CT) — Undergo chest CT
  Other Names: Undergo chest CT
Other: Laboratory Biomarker — Correlative studies

SUMMARY:
This research trial studies the long term follow-up for early detection of lung cancer in current or former smokers. Following up on smokers by collecting and analyzing specimens in the laboratory, performing chest computed tomography (CT) scans, as well as reviewing medical records may help doctors detect lung cancer at an earlier stage.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide screening for lung cancer in an underserved and high risk population for lung cancer.

II. To collect clinical and demographic information and research bio specimens prospectively on high risk individuals.

III. To analyze the association between suspected lung cancer risk factors and outcomes such as pre-malignant lesions and diagnosis of lung cancer.

IV. To identify and validate biomarkers that are associated with lung cancer risk factors and premalignant lesions.

V. To assess the association between patient characteristics and test results to the genetic and histological characteristics of lung preinvasive lesions and cancers.

VI. To describe this high-risk cohort and to identify the patients eligible for future clinical trials (e.g. chemoprevention).

OUTLINE:

Patients are followed up at 1, 2, 3, 4, and 5 years and undergo collection of sputum, nasal epithelium, buccal epithelium, blood, and urine samples. Patients also undergo pulmonary function tests, chest CT, and review of medical records.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker or former smoker, if former smoker participants must have quit smoking within the past 15 years
* >= 30 pack year of smoking history
* Participant is uninsured

Exclusion Criteria:

* History of diagnosis/treatment of lung cancer in the past 2 years
* History of head/neck or esophageal cancer in the last 1 year
* Inability to provide informed consent

Ages: 55 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Current or former smokers
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Candidate biomarkers of risk or of early diagnosis | Up to 5 years.
  Will validate the performance of the candidate biomarkers of risk or of early diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grogan, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided